CLINICAL TRIAL: NCT02149901
Title: Effect of Drinking Water on the Pressor Response to Pseudoephedrine in Patients With Autonomic Failure
Brief Title: Water and Sudafed in Autonomic Failure
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: funding terminated
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Emily M. Garland, Research Associate Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 140547; P01HL056693 (NIH); UL1TR000445 (NIH)
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Shy-Drager Syndrome; Multiple System Atrophy
Keywords: Pure Autonomic Failure; Multiple System Atrophy; Pseudoephedrine; Water; Osmopressor
MeSH Terms: conditions — Shy-Drager Syndrome; Multiple System Atrophy; Pure Autonomic Failure | interventions — Pseudoephedrine; Water; Drinking Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pseudoephedrine + 480 ml water (Experimental): Pseudoephedrine 30 mg PO 45 minutes before water 480 ml
  Interventions: Drug: Pseudoephedrine + 480 ml water
- Pseudoephedrine + 50 ml water (Placebo Comparator): Pseudoephedrine 30 mg PO 45 minutes before water 50 ml
  Interventions: Drug: Pseudoephedrine + 50 ml water
- Placebo + 480 ml water (optional) (Experimental): Placebo PO 45 minutes before water 480 ml
  Interventions: Other: Placebo + 480 ml water (optional)
- Placebo + 50 ml water (optional) (Placebo Comparator): Placebo PO 45 minutes before water 50 ml
  Interventions: Other: Placebo + 50 ml water (optional)

INTERVENTIONS:
Drug: Pseudoephedrine + 480 ml water — 30 mg pseudoephedrine to be given with a pressor dose (480 ml) of drinking water
  Other Names: Sudafed; drinking water
  Arms: Pseudoephedrine + 480 ml water
Drug: Pseudoephedrine + 50 ml water — Pseudoephedrine given with a non-pressor (50 ml) dose of drinking water
  Other Names: Sudafed; drinking water
  Arms: Pseudoephedrine + 50 ml water
Other: Placebo + 480 ml water (optional) — placebo PO with a pressor (480 ml) dose of drinking water
  Other Names: drinking water
  Arms: Placebo + 480 ml water (optional)
Other: Placebo + 50 ml water (optional) — placebo PO with a non-pressor (50 ml) dose of drinking water
  Other Names: drinking water
  Arms: Placebo + 50 ml water (optional)

SUMMARY:
The specific aim of this study is to determine whether water ingestion potentiates the pressor response to pseudoephedrine in patients with primary disorders of autonomic failure. The study design will enable us to also evaluate the pressor response to water alone and to pseudoephedrine alone. In a secondary analysis, we will compare the results in patients with two autonomic disorders, pure autonomic failure (PAF) and multiple system atrophy (MSA). We hypothesize that drinking water following a dose of pseudoephedrine will lead to a greater increase in blood pressure than pseudoephedrine alone.

DETAILED DESCRIPTION:
The maximal pressor response to water is reached when other pressor agents are only beginning to act. In addition to the therapeutic value of water ingestion alone, the blood pressure-raising effects of agents that increase sympathetic nervous system tone, such as phenylpropanolamine, are potentiated by water drinking. These drug interaction effects can be exploited in the treatment of orthostatic hypotension with the combination of water and a sympathomimetic potentially able to increase blood pressure to a greater extent and for a longer period of time than either water or the medication alone. However, the interaction can also lead to potentially dangerous blood pressure surges.

This protocol requires an initial screening history and physical of study participants, including safety labs and EKGs, and evaluation of their autonomic nervous system status following the consent process. If the patient meets study criteria and is willing to undergo study testing, the 4-way crossover protocol will follow.

Study Testing days 1 and 2 Arm 1: Pseudoephedrine 30 mg PO + 50 ml water Arm 2: Pseudoephedrine 30 mg PO + 480 ml water

* Testing will be performed at the same time of day for all studies, at least 2 hours after a meal to avoid any confounding effects from postprandial hypotension.
* A saline lock will be inserted for blood sampling at least 30 minutes before baseline data collection.
* Participants will be asked to empty their bladders before beginning the test to avoid any effect of a full urinary bladder on peripheral sympathetic activity.
* Participants will be seated comfortably in a chair. They will be asked to remain in the seated position for the duration of the study.
* The Dinamap electrocardiographic and blood pressure (brachial cuff) recorder will be attached to the patient and set up for measurements every 5 minutes throughout the study with digital download into the ADC (Autonomic Dysfunction Center) BP database.
* Participants will also be instrumented with EKG, finger cuff and sensor for continuous monitoring of blood pressure, heart rate, respiration, SpO2, stroke volume, systemic vascular resistance, and cardiac output, using a Nexfin system and Ivy Biomedical Vital-Guard monitor.
* After a 30 minute baseline monitoring period (time -30 min to 0 min), 4 ½ teaspoons of blood will be collected for osmolality measurement and assays of hormones that regulate blood pressure.
* The subject will then be given 30 mg of pseudoephedrine PO (time 0 min). Monitoring will be continued for 45 minutes.
* At 45 minutes, the participant will be asked to drink 50 ml (Arm 1) or 480 ml (Arm 2) of water.
* Additional blood samples (4 ½ teaspoons) for osmolality and BP-regulating hormones will be collected 30 and 60 minutes after water (+75 and +105 minutes of study).
* Monitoring will be continued until + 135 min.
* At 135 minutes, the study will end for the day. The timing of pseudoephedrine administration relative to water ingestion and the duration of the monitoring period are based on previous results3 and pharmacokinetic data7 reporting a Tmax for pseudoephedrine between 1 and 2 hours. Testing on study day 2 will be identical with the participant consuming the alternate water volume.

Study Testing days 3 and 4 are optional Arm 3: Placebo PO + 50 ml water Arm 4: Placebo PO + 480 ml water Testing will be performed according to the same schedule as for Arms 1 and 2. Instrumentation will be limited to the Dinamap electrocardiographic and blood pressure (brachial cuff) recorder set up for measurements every 5 minutes throughout the study for Arms 3 and 4.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years, with
* Neurogenic orthostatic hypotension, ≥30 mmHg drop in SBP within 5 minutes of standing,
* Associated with impaired autonomic reflexes, as determined by absence of blood pressure overshoot during phase IV of the valsalva maneuver,
* Absence of other identifiable causes of autonomic neuropathy, and
* Able and willing to provide informed consent

Exclusion Criteria

* Pregnancy
* Current smoking habit
* Systemic illnesses known to produce autonomic neuropathy, including but not limited to diabetes mellitus, amyloidosis, monoclonal gammopathy of unknown significance, and autoimmune neuropathies.
* Known intolerance to pseudoephedrine
* Pre-existing sustained severe hypertension (BP > 180/110 mmHg in the sitting position)
* Clinically unstable coronary artery disease or major cardiovascular or neurological event in the past 6 months.
* Any other significant systemic, hepatic, cardiac or renal illness
* Use of MAO-I (i.e. selegiline; rasagiline - Azilect, linezolid and others) within 14 days
* Known closed-angle glaucoma
* Clinically meaningful arrhythmias
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies or an unpredictable schedule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure in each Aim will be the peak increase in systolic blood pressure after pseudoephedrine or placebo relative to baseline (delta SBP). | between 60 and 120 minutes after pseudoephedrine or placebo

SECONDARY OUTCOMES:
Change in diastolic blood pressure relative to baseline | between 60 and 120 minutes after pseudoephedrine or placebo
Change in heart rate relative to baseline | between 60 and 120 minutes after pseudoephedrine or placebo
Absolute systolic blood pressure after treatment | between 60 and 120 minutes after pseudoephedrine and placebo
Absolute diastolic blood pressure after treatment | between 60 and 120 minutes after pseudoephedrine or placebo
area under the curve for systolic blood pressure from baseline to 135 minutes post-treatment | from baseline to 135 minutes after pseudoephedrine or placebo
  Area under the curve can better measure an extension of the duration of response.
Peak plasma norepinephrine concentration after treatment | between baseline and 135 minutes after pseudoephedrine or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Emily M Garland, PhD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Jordan J, Shannon JR, Grogan E, Biaggioni I, Robertson D. A potent pressor response elicited by drinking water. Lancet. 1999 Feb 27;353(9154):723. doi: 10.1016/S0140-6736(99)99015-3. No abstract available. PMID 10073520
- [Background] Jordan J, Shannon JR, Black BK, Ali Y, Farley M, Costa F, Diedrich A, Robertson RM, Biaggioni I, Robertson D. The pressor response to water drinking in humans : a sympathetic reflex? Circulation. 2000 Feb 8;101(5):504-9. doi: 10.1161/01.cir.101.5.504. PMID 10662747
- [Background] Jordan J, Shannon JR, Diedrich A, Black B, Robertson D, Biaggioni I. Water potentiates the pressor effect of ephedra alkaloids. Circulation. 2004 Apr 20;109(15):1823-5. doi: 10.1161/01.CIR.0000126283.99195.37. Epub 2004 Apr 5. PMID 15066944
- [Background] Kobayashi S, Endou M, Sakuraya F, Matsuda N, Zhang XH, Azuma M, Echigo N, Kemmotsu O, Hattori Y, Gando S. The sympathomimetic actions of l-ephedrine and d-pseudoephedrine: direct receptor activation or norepinephrine release? Anesth Analg. 2003 Nov;97(5):1239-1245. doi: 10.1213/01.ANE.0000092917.96558.3C. PMID 14570629
- [Background] Rothman RB, Vu N, Partilla JS, Roth BL, Hufeisen SJ, Compton-Toth BA, Birkes J, Young R, Glennon RA. In vitro characterization of ephedrine-related stereoisomers at biogenic amine transporters and the receptorome reveals selective actions as norepinephrine transporter substrates. J Pharmacol Exp Ther. 2003 Oct;307(1):138-45. doi: 10.1124/jpet.103.053975. Epub 2003 Sep 3. PMID 12954796
- [Background] Lu CC, Diedrich A, Tung CS, Paranjape SY, Harris PA, Byrne DW, Jordan J, Robertson D. Water ingestion as prophylaxis against syncope. Circulation. 2003 Nov 25;108(21):2660-5. doi: 10.1161/01.CIR.0000101966.24899.CB. Epub 2003 Nov 17. PMID 14623807
- [Background] Kanfer I, Dowse R, Vuma V. Pharmacokinetics of oral decongestants. Pharmacotherapy. 1993 Nov-Dec;13(6 Pt 2):116S-128S; discussion 143S-146S. PMID 7507589
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations. A review and computer program. Control Clin Trials. 1990 Apr;11(2):116-28. doi: 10.1016/0197-2456(90)90005-m. PMID 2161310